CLINICAL TRIAL: NCT07030777
Title: The Experience of Giving Birth With Remifentanil for Pain Relief: A Qualitative Study of Mothers and Midwives
Status: Recruiting | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Principal Investigator, Patricia Duch, M.D. Consultant, obstetric anaesthetist, Nordsjaellands Hospital
Other Study IDs: 103
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Pain Management in Pregnant Women; Remifentanil; Midwife; Qualitative Research; Birth; Labour Analgesia
Keywords: Labour analgesia; remifentanil for labour analgesia; qualitative research; midwifes experiences with remifentanil; giving birth with remifentanil

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Midwifes: Group 1: Midwives This group includes licensed midwives who have administered remifentanil for pain relief during labor. Participants will be interviewed about their experiences with providing care during remifentanil-supported childbirth, including perceptions of efficacy, safety, and clinical workflow.
- Laboring Women: Group 2: Laboring Women This group consists of women who gave birth using remifentanil patient-controlled analgesia (PCA) for pain relief during labor. Participants will be interviewed about their lived experience of pain management, decision-making, and overall birth experience using remifentanil.

SUMMARY:
Background:

Remifentanil is an ultra-short-acting opioid used for labor pain relief in several countries, offering stronger analgesia than nitrous oxide but less than epidural anesthesia. While internationally established, remifentanil has not yet been implemented in Denmark.

Objective:

This study aims to explore and deepen our understanding of the childbirth experience with remifentanil for pain relief, from both the birthing woman's and the midwife's perspectives.

Methods:

A qualitative study based on interviews with women who gave birth using remifentanil and the midwives involved in their care.

DETAILED DESCRIPTION:
Background:Remifentanil is an ultra-short-acting opioid used for labor pain relief in several countries, offering stronger analgesia than nitrous oxide but less than epidural anesthesia. While internationally established, remifentanil has not yet been implemented in Denmark. Objective:This study aims to explore and deepen our understanding of the childbirth experience with remifentanil for pain relief, from both the birthing woman's and the midwife's perspectives. Methods: A qualitative study based on semi-structured interviews with women who gave birth using remifentanil and the midwives involved in their care. The analysis will be a thematic content analysis. All Danish or English speaking labouring women and midwifes at North Zealand hospital giving birth/attending birth with remifentanil for labour pain are eligible to be included during the study period. After written consent the interview will be conducted 4-10 days after the birth.

ELIGIBILITY:
Inclusion Criteria:

1. Women in labor aged 18 years or older who receive remifentanil for pain relief during childbirth at the labor ward in Hillerød.
2. Midwives who participate in childbirths where remifentanil is used as pain relief.

Exclusion Criteria

1)Women in labor who do not speak Danish or English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — People experiencing labor pain
Study Population: Study Population and Recruitment Setting Participants will be initially approached during their hospital admission after giving birth using remifentanil for labor analgesia at the labor ward in Hillerød. At this point, they will receive verbal and written information about the study and may be included if they provide informed consent.
  Midwives will be contacted after the relevant birth has taken place. They will be informed about the study and included if they agree to participate.
  If the mother and/or midwife consents to participate, they will be contacted by phone to schedule a semi-structured interview 4-10 days postpartum
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Experiential understanding of remifentanil-assisted labor from the perspectives of mothers | Interviews conducted within 4-10 days postpartum
  The co-primary outcome is the in-depth qualitative description of how women experience the use of remifentanil for labor pain relief. The outcome will be derived through thematic analysis of semi-structured interview data, aiming to identify key themes related to pain relief, side-effects, safety, communication, autonomy, and overall birth experience. No quantitative scale will be used.
Experiential understanding of remifentanil-assisted labor from the perspectives of midwives | Time Frame: Interviews conducted within 4-10 days postpartum
  Description: The co-primary outcome is the in-depth qualitative description of how midwifes experience the use of remifentanil for labor pain relief. The outcome will be derived through thematic analysis of semi-structured interview data, aiming to identify key themes related to pain relief, side-effects, safety, communication, autonomy, and overall birth experience. No quantitative scale will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Duch, MD, Study Chair — Department of Anaesthesia, Copenhagen University Hospital, North Zealand, Hillerød, Denmark
Locations (3):
- Denmark (3):
  - University Hospital of Copenhagen, North Zealand Hospital, Hillerød, Select State
  - Department of Anaesthesia and Intensive care, University Hospital of Southern Denmark, Kolding, Denmark, Kolding
  - Præhospital center, Næstved

IPD SHARING:
Plan to Share IPD: Yes
IPD Sharing Statement Individual participant data (IPD) in the form of full interview transcripts will not be shared due to privacy concerns and the qualitative, sensitive nature of the material. However, de-identified quotes and aggregated thematic analysis results may be shared as part of the published findings or upon reasonable request for academic purposes, in accordance with participants' consent and ethical approval.